CLINICAL TRIAL: NCT04881877
Title: A Functional Performance and Acceptability Study of a Synthetic Nitrile Male Condom, and a Latex Graphene Male Condom Compared to a Standard Latex Male Condom
Brief Title: Functional Performance and Acceptability Study of Synthetic Nitrile, and Latex Graphene, Compared to Standard Latex Male Condom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Mags Beksinska (Other)
Responsible Party: Sponsor-Investigator, Prof Mags Beksinska, Deputy Executive Director, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Karex
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Functional Performance
Keywords: synthetic nitrile male condom; latex graphene male condom; latex male condom

STUDY DESIGN:
Intervention Model Description: The study is a randomized cross-over trial to evaluate the functional performance of two new male condoms compared to a control latex male condom.
Who Masked: Outcomes Assessor
Masking Description: Analysts will be blinded until all data have been captured and the primary analysis programs have been verified. Likewise, all reasonable attempts will be made to keep other non-monitor staff blinded during the course of the study. The statistician analyzing the data will not be blinded. Due to slight differences related to colour of the study products, it will not be possible to blind participants and clinic staff associated with the project
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Synthetic nitrite Condom (Experimental): Participants will be randomized to condom use order. Participants will be provided with 5 synthetic nitrite condoms at the first visit and switched to 5 of either the latex graphene condom or latex condom at visit 2 and 3. All couples will use each of the 3 condom types during the study
  Interventions: Device: Synthetic nitrite Condom; Device: Latex and graphene Condom; Device: Standard latex condom
- Latex and graphene Condom (Experimental): Participants will be randomized to condom use order. Participants will be provided with 5 latex graphene condoms at the first visit and switched to 5 of either the synthetic nitrite condom or latex condom at visit 2 and 3. All couples will use each of the 3 condom types during the study.
  Interventions: Device: Synthetic nitrite Condom; Device: Latex and graphene Condom; Device: Standard latex condom
- Standard latex condom: (Experimental): Participants will be randomized to condom use order. Participants will be provided with 5 latex condom at the first visit and switched to 5 of either the latex graphene condom or synthetic nitrite condoms at visit 2 and 3. All couples will use each of the 3 condom types during the study.
  Interventions: Device: Synthetic nitrite Condom; Device: Latex and graphene Condom; Device: Standard latex condom

INTERVENTIONS:
Device: Synthetic nitrite Condom — The condoms is composed of a synthetic nitrile rubber latex and 170 mm in length and is 53mm wide. It has a teat ended shape and bead retention mechanism at the top. It is pre-lubricated with silicone oil. It has a shelf-life of 5 years and clear and colourless. It is manufactured by Karex Industries. It is currently experimental.
Device: Latex and graphene Condom — The condom is composed of a natural rubber latex with graphene. It is 170 mm in length and is 53mm wide. It has a teat ended shape and bead retention mechanism at the top. It is pre-lubricated with silicone oil. It has a shelf-life of 5 years and is greyish in colour. It is manufactured by Karex Industries. It is currently experimental.
Device: Standard latex condom — The condoms is composed of a natural rubber latex. It is 180 mm in length and is 53mm wide. It has a teat ended shape and bead retention mechanism at the top. It is pre-lubricated with silicone oil. It has a shelf-life of 5 years and is natural in colour. It is manufactured by Karex Industries. It has World Health Organisation (WHO)/UNFPA, India Drug Control Authority, Conformitè Europëenne (CE) Mark of the European Union, South African Bureau of Standards and US FDA approval

SUMMARY:
Two new male condoms have been developed - one made of synthetic nitrile and the other made of latex graphene. Both new condoms are of the same design as a standard latex male condom. The aim of this study is to evaluate the functional performance of two new male condoms compared to a control latex male condom. Couples enrolled in the study will be asked to use five latex graphene, five synthetic nitrile and five latex male condoms in a randomized type order. Function, safety, and acceptability will be assessed at three follow-up visits approximately one month apart after enrolment.

DETAILED DESCRIPTION:
Two new male condoms have been developed - one made of synthetic nitrile and the other made of latex graphene. Both new condoms are of the same design as a standard latex male condom.

Purpose: The aim of the study is to evaluate the functional performance of two new male condoms compared to a control latex male condom.

Study design: The study is a randomized three-period cross-over trial of two new male condoms and a control latex male condom. The study will enrol 240 couples, anticipating that at least 200 couples will complete the study. Each couple will be asked to use five latex graphene, five synthetic nitrile and five latex male condoms in a randomized type order. Function, safety, and acceptability will be assessed at three follow-up visits approximately one month apart after enrolment. Couples will complete a Condom Log at their homes which gathers data on experience after use of each condom.

Primary Objective: To ascertain the functional performance of a latex graphene and a synthetic nitrile compared to a control latex male condom. Primary endpoints will be total clinical failure and total condom failure.

Secondary Objectives: Acceptability and safety data (as determined by the number of adverse events) occurring with each male condom type.

Population: The target population will be 240 urban, sexually-active couples who are experienced users of male condoms. Recruitment will be from the Commercial City MatCH Research Unit (MRU) site and other workplace sites in the eThekwini District.

Men and women will be told about the study. If a man/woman expresses interest in participating, they will be given the study information sheet to read, which will describe the study requirements and their potential role/partners potential in the study. If they agree to take part in the research, they will be asked to give the information sheet to their partner. If both partners in the couple are willing to participate, they will be invited to visit the enrolment site or the MRU Commercial City site and asked to provide written informed consent. Both partners will be screened to ensure they meet the requirements for study participation.

A physical examination will be undertaken to exclude visible symptoms of sexually transmitted infections. If symptoms are observed the participant will be referred to a Department of Health clinic or their doctor for treatment. A urine pregnancy test will be conducted at screening to exclude pregnancy. Both partners in the couple will need to provide the study with a copy of HIV results which are not older than 2 months. If HIV testing results are not available, voluntary HIV counselling and testing will be offered and conducted by study staff.

The consent process and all checklists, condom use logs and surveys used in the research will be written and conducted in a language that is understandable to the participant, and all relevant documents will be translated into isiZulu. Enrolled participants will be asked to use five latex graphene, five synthetic nitrile and five latex male condoms. They will be asked to return for follow-up after using five of each type of device.

At enrolment, baseline data will be gathered on participant demographics and past male condom use via the baseline questionnaire using a dildo model, the study staff will demonstrate male condom fitting and train the participants in the proper use of their first assigned male condom. Further, they will re-emphasize the instructions on how to complete the condom use log. Couples will be given one condom log to complete together. Couples will be told that they do not have to use the study male condoms during consecutive acts of intercourse. They will also be counselled on Pre Exposure Prophylaxis (PrEP) and referred to a local facility that provides PrEP should they wish to initiate PrEP. The study staff will discuss with the couple an approximate timeframe for use of all five condoms and a suitable follow-up date will be scheduled. This date will be noted on an appointment slip. Couples will be encouraged to come back if their condoms are finished before the due date and will be given the research study contact details to call for any appointment changes.

During the first follow-up visit, couples will be interviewed about their first assigned condom type and they will receive their next condom packet within their second assigned (randomized) use sequence. In the second follow-up visit, couples will be interviewed about their second assigned condom type and they will receive their next condom packet within their third assigned (randomized) use sequence.

In the third follow-up visit, couples will be interviewed about their third assigned condom type and will be discontinued from study participation. Data on device function, safety and acceptability for each condom type will be collected during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

All couples enrolled in this research must meet the following selection criteria:

1. Be between the ages of 18 and 45 years (inclusive);
2. Be literate (able to read a newspaper or letter easily);
3. Have been in an exclusive (monogamous) sexual relationship with partner for at least 6 months; and intend to continue to be an exclusive (monogamous) sexual relationship with partner with their spouse or partner while participating in this research study;
4. Not planning a pregnancy during the time of the research study;
5. Be sexually active (defined as having at least two vaginal coital acts per week and not being abstinent in the month prior to enrolment);
6. Not have any genital piercings, use genital beading or any other drugs or non-study devices that can affect sexual performance;
7. Not have known sensitivities or allergies to latex, polyurethane, vaginal/sexual lubricants or the lubricants used on condoms;
8. Be without observable evidence of Sexually transmitted infections (STI) as determined through syndromic diagnosis and vaginal/penile examination;
9. Not be HIV positive
10. Willing to give informed consent;
11. Willing to complete the male condom coital use logs;
12. Willing to use the study condoms as directed;
13. Willing to adhere to the follow-up schedule and all study procedures;
14. Willing to provide research study staff with an address, phone number or other locator information while participating in the study; and,
15. Willing to participate in the study for the duration of 15 condom uses (approximately 3- 5 months.
16. Willing to have fingerprint scan to check for co-enrolment in other research projects Female partner only: -
17. Using hormonal or other non-barrier contraception (e.g. Oral Contraceptives (OC), injectable, implant, Intra Uterine Device (IUD), or have had a tubal sterilization);
18. Must not be pregnant (as determined by pregnancy testing)
19. Not be menopausal (defined as 12 months without menstruation);
20. Not have had a hysterectomy; Male partner only: -
21. Not have known erectile or ejaculatory dysfunction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Clinical breakage | 3-5 months
  Clinical breakage is defined as breakage during sexual intercourse or during withdrawal of the male condom from the vagina. Clinical breakage is breakage with potential adverse clinical consequences. The clinical breakage rate is calculated by dividing the number of male condoms reported to have broken during sexual intercourse or during withdrawal by the number of male condoms used during sexual intercourse.
Non-Clinical breakage | 3-5 months
  Defined as breakage noticed before sexual intercourse or occurring after withdrawal of the male condom from the vagina. Non-clinical breakage is breakage with no potential adverse clinical consequences. The non-clinical breakage rate is calculated by dividing the number of male condoms reported to have broken before sexual intercourse or after withdrawal by the number of male condom packages opened
Total breakage | 3-5 months
  Total breakage is defined as the sum of all male condom breakages at any time before, during or after sexual intercourse. It includes both clinical breakages and non-clinical breakages. The total breakage rate is calculated by dividing the total number of male condoms that broke by the number of male condom packages opened.
Slippage | 3-5 months
  Slippage is defined as an instance when a male condom slips completely off the penis during sexual intercourse or during withdrawal from the vagina. The slippage rate is calculated by dividing the number of male condoms that slipped by the number of male condoms used during sexual intercourse.
Total clinical failure | 3-5 months
  Total clinical failure is defined as the sum of male condoms that clinically break or slip, or any additional failure modes(s) identified in the risk assessment which results in the reduction of the male condom protective function. The total clinical failure rate is calculated by dividing the number of male condoms with a clinical failure by the number of male condoms used during sexual intercourse.
Total male condom failure | 3-5 months
  Total male condom failure is defined as a male condom for which a non-clinical breakage, clinical breakage or slippage occurs, or is associated with any additional failure modes(s) identified in the risk assessment. The male condom failure rate is calculated by dividing the number of male condoms that fail by the number of male condom packages opened

SECONDARY OUTCOMES:
Safety assessed by genitourinary adverse events | 3-5 months
  Proportion of participants with symptoms of and proportion of male condom uses with reports of genitourinary irritation during or immediately after any of the five separate uses will be calculated. Medical and serious adverse events will be classified by relatedness, expectedness and severity
Acceptability assessed by the frequency of key acceptability endpoints | 3-5 months
  Frequency of key acceptability endpoints will be calculated and include: comfort in use; ease of insertion and removal; like or dislike of product attributes; adequacy and feel of lubrication and sensitivity and stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Mags Beksinska, PhD, Study Director — MatCH Research Unit [Maternal, Adolescent and Child Health Research Unit]
Locations (1):
- MatCH Research Unit [Maternal, Adolescent and Child Health Research Unit], Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warren M. Condoms: the multipurpose prevention technologies that already exist. BJOG. 2014 Oct;121(Suppl 5):9-11. doi: 10.1111/1471-0528.12913. No abstract available. PMID 25335833
- [Background] Martinez G, Copen CE, Abma JC. Teenagers in the United States: sexual activity, contraceptive use, and childbearing, 2006-2010 national survey of family growth. Vital Health Stat 23. 2011 Oct;(31):1-35. PMID 22256688
- [Background] World Health Organization Department of Reproductive Health and Research (WHO/RHR), John Hopkins Bloomberg School of Public Health/Center for Communication Programs (CCP). Family Planning: A Global Handbook for Providers (2018 update) [Internet]. Baltimore and Geneva: CCP and WHO; 2018 [CITED 2019 June 20]. 442p. Available from http://apps.who.int/iris/bitstream/10665/260156/1/9780999203705- eng.pdf?ua=1.
- [Background] UNFPA, Universal access to Reproductive Health: Progress and Challenges. https://www.unfpa.org/sites/default/files/pubpdf/UNFPA_Reproductive_Paper_20160120_online.pdf
- [Background] Shisana O, Rehle T, Simbayi LC, et al. South African national HIV prevalence, incidence, behaviour and communication survey 2017: Health and wellbeing: Human Science Research Council Press; 2017.
- [Background] Muchiri E, Odimegwu E, DeWet N. HIV risk perception and consistency in condom use among adolescents and young adults in urban Cape Town, South Africa: a cumulative risk analysis. S Afr J Infect Dis [Internet]. 2017 [cited 2019 Sep 8]; 32(3):105-110. Available from: https://doi.org/10.1080/23120053.2017.1332800
- [Background] Beksinska M, Wong R, Smit J. Male and female condoms: Their key role in pregnancy and STI/HIV prevention. Best Pract Res Clin Obstet Gynaecol. 2020 Jul;66:55-67. doi: 10.1016/j.bpobgyn.2019.12.001. Epub 2019 Dec 14. PMID 32007451
- [Background] Pumphrey RS. Allergy to Hevea latex. Clin Exp Immunol. 1994 Dec;98(3):358-60. doi: 10.1111/j.1365-2249.1994.tb05497.x. No abstract available. PMID 7994899
- [Background] Bousquet J, Flahault A, Vandenplas O, Ameille J, Duron JJ, Pecquet C, Chevrie K, Annesi-Maesano I. Natural rubber latex allergy among health care workers: a systematic review of the evidence. J Allergy Clin Immunol. 2006 Aug;118(2):447-54. doi: 10.1016/j.jaci.2006.03.048. Epub 2006 Jul 3. PMID 16890771
- [Background] Walsh TL, Frezieres RG, Peacock K, Nelson AL, Clark VA, Bernstein L. Evaluation of the efficacy of a nonlatex condom: results from a randomized, controlled clinical trial. Perspect Sex Reprod Health. 2003 Mar-Apr;35(2):79-86. PMID 12729137
- [Background] Gallo MF, Grimes DA, Lopez LM, Schulz KF. Non-latex versus latex male condoms for contraception. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD003550. doi: 10.1002/14651858.CD003550.pub2. PMID 16437459
- [Background] George G, Sisupal SB, Tomy T, Pottammal BA, Kumaran A, Suvekbala V, Gopimohan R, Sivaram S, Ragupathy L. Thermally conductive thin films derived from defect free graphene-natural rubber latex nanocomposite: Preparation and properties. Carbon N Y. 2017 Aug;119:527-534. doi: 10.1016/j.carbon.2017.04.068. PMID 28775386
- [Background] ISO 29943-1:2017 Condoms - Guidance on clinical studies - Part 1: Male condoms, clinical function studies based on self-reports. https://www.iso.org/standard/62497.html
- [Background] Steiner M, Piedrahita C, Joanis C, Glover L, Spruyt A. Condom Breakage and Slippage Rates Among Study Participants in Eight Countries. Int Fam Plan perspect 1994 ;20:55-58